CLINICAL TRIAL: NCT05275036
Title: Assessment of Early-detection Based on Liquid Biopsy in Lymphoid Malignancies: a Multi-center Prospective Observational Study
Brief Title: Assessment of Early-detection Based on Liquid Biopsy in Lymphoid Malignancies
Acronym: ASCEND-LYM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Huiqiang Huang, chief physician, Sun Yat-sen University
Other Study IDs: BRCD2022003
Record Dates: First submitted 2022-02-28; First posted 2022-03-11 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Lymphoma
Keywords: lymphoma, early detection, liquid biopsy
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, white blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Arm: Participants with new diagnosis of lymphoid malignancies, from whom blood samples will be collected.
  Interventions: Device: early detection test
- Benign Arm: Participants with new diagnosis of benign lymphoid diseases, from whom blood samples will be collected.
  Interventions: Device: early detection test

INTERVENTIONS:
Device: early detection test — Blood collection and early detection testing

SUMMARY:
ASCEND-LYM is a prospective, multi-center, observational study aimed at detecting early stage lymphoma and constrcuting prognostic model by combined assays of cfDNA methylation and other biomarkers. The study will enroll approximately 493 participants including lymphoid malignancies and benign diseases.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Age 40-75 years at the day of consenting to the study.
* Able to provide a written informed consent.

Additional Inclusion Criteria for Cancer Participants:

* No prior cancer treatment (local or systematic) prior to blood draw.
* High suspicious or pathologically confirmed lymphoid malignancies within 42 days prior to blood draw.

Additional Inclusion Criteria for Benign Disease Participants:

* No prior radical treatment of the benign diseases prior to study blood draw
* Pathologically confirmed diagnosis of lymphoid benign diseases within 90 days prior to blood draw.

Exclusion Criteria for All Participants:

* Insufficient qualified blood samples.
* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 7 days prior to blood draw.
* Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw, such as rheumatic drugs (methotrexate, cyclophosphamide, or azathioprine), or endocrine drugs (tamoxifen).

Additional Exclusion Criteria for Cancer Participants:

* With other known malignant tumors or multiple primary tumors.
* Lymphoid malignancies unable to comfirmed by imaging tests or pathological cancer diagnosis within 42 days after the blood draw.

Additional Exclusion Criteria for Benign Disease Participants:

* With other known malignant tumors or comfirmed lymphoid malignancies.
* Lymphoid benign diseases unable to comfirmed by imaging tests or pathological cancer diagnosis within 42 days after the blood draw.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from the participating medical center and assigned into two arms, including participants with new diagnosis of lymphoid malignancies and benign lymphoid diseases.
Sampling Method: Non-Probability Sample
Enrollment: 493 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of early detection model for lymphoma based on cfDNA methylation or combined with other biomarkers. | 12 months

SECONDARY OUTCOMES:
The sensitivity and specificity of the optimal model in lymphoma patients at different clinical stages. | 12 months
The sensitivity and specificity of the optimal model in different subtypes of lymphoma patients. | 12 months
The rate of high-risk patients found by prognostic model for lymphoma based on cfDNA methylation or combined with other biomarkers. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Ph.D, Principal Investigator — Department of Medical Oncology, Sun Yat-sen University Cancer Center
Locations (1):
- SunYat-sen university cancer center, Guangzhou, China